CLINICAL TRIAL: NCT03430453
Title: Observational Study : Minimal Intensity of Stimulation During Ultrasound Guided Peripheral Nerve Block According to Anatomic Needle Type Position
Brief Title: Monitoring of Intensity of Stimulation and Injection Pressure in US Guided Peripheral Nerve Block According to Anatomic Needle Type Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF8924
Record Dates: First submitted 2015-09-22; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2015-09

CONDITIONS: Orthopedic Surgery
Keywords: Regional Anesthesia; Ultrasound guidance; Nerve stimulation; Orthopedic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with ultrasound guided peripheral nerve blockade (Experimental): A needle is placed at the target under ultrasound guidance, the nerve stimulator is turned on and the intensity increased until motor response is observed.
  Interventions: Procedure: Measure of the minimal intensity of stimulation during ultrasound guided peripheral nerve blockade

INTERVENTIONS:
Procedure: Measure of the minimal intensity of stimulation during ultrasound guided peripheral nerve blockade — A needle is placed at the target under ultrasound guidance, the nerve stimulator is turned on and the intensity increased until motor response is observed. The Minimal Intensity of Stimulation is recorded before injection of local anesthetic

SUMMARY:
The purpose of the study is define the minimal intensity of stimulation range at which the needle is closed to the nerve without penetrating its surface (epineurium layer) in ultrasound guided peripheral nerve blockade

DETAILED DESCRIPTION:
The needle is placed at the target under ultrasound guidance the nerve stimulator is turned on and the intensity increased until motor response is observed the Minimum Intensity Observation (MIS) is recorded before injection of local anesthetic

ELIGIBILITY:
Inclusion Criteria:

* Patient who need a Orthopedic surgery
* Peripheral nerve block
* More or equal to 18 years old
* I to III ASA classification status
* Benefit from an insurance regimen

Exclusion Criteria:

* severe coagulopathy
* allergy to local anesthetics
* local cutaneous lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of Minimum Intensity Stimulation | estimated between 2 minutes and 20 minutes.
  Minimal Intensity Stimulation (MIS) was measured Using a specific nerve stimulator (modified HNS 12 B. BRAUN, Melsungen, Germany) ; the value are noted in mA. [0- 1.5].
  The time frame is only related to procedure of PNB. In other term, the period of assessment should be estimated between 2 minutes and 20 minutes.

SECONDARY OUTCOMES:
tissure pressure at the target | estimated between 2 minutes and 20 minutes.
  Tissue pressure at the target was measured Using a specific pressure sensor (compuflow pump Milestone Scientific, Livingston, NJ, USA) ; the value are noted in mm Hg. [0- 900].
  from beginning to end of ultrasound guided peripheral nerve blockade

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - University Hospital of Annecy, Annecy
  - University hospital of Bordeaux, Bordeaux
  - University hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Colmar, Colmar
  - University hospital of limoges, Limoges
  - University hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University hospital of Nice, Nice
  - University Hospital of Reims, Reims

REFERENCES:
- [Derived] Varobieff M, Choquet O, Swisser F, Coudray A, Menace C, Molinari N, Bringuier S, Capdevila X. Real-Time Injection Pressure Sensing and Minimal Intensity Stimulation Combination During Ultrasound-Guided Peripheral Nerve Blocks: An Exploratory Observational Trial. Anesth Analg. 2021 Feb 1;132(2):556-565. doi: 10.1213/ANE.0000000000005308. PMID 33323786
- [Derived] Capdevila M, Choquet O, Saporito A, Djanikian F, Swisser F, Marques M, Bringuier S, Capdevila X. Injection pressure monitoring during peripheral nerve blocks: from bench to operating theatre. Anaesth Crit Care Pain Med. 2020 Oct;39(5):603-610. doi: 10.1016/j.accpm.2020.03.022. Epub 2020 Aug 10. PMID 32791158